CLINICAL TRIAL: NCT01433237
Title: A Retrospective Study on the Diagnostic Value of Serum miR-206 in Rhabdomyosarcoma
Brief Title: Studying Biomarkers in Samples From Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B1; COG-ARST12B1 (Other: Children's Oncology Group); ARST12B1 (Other: Children's Oncology Group); NCI-2011-03457 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; adult rhabdomyosarcoma; alveolar childhood rhabdomyosarcoma; adult soft tissue sarcoma; childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma; Rhabdomyosarcoma | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether circulating muscle-specific microRNAs, especially serum miR-206, are potential biomarkers for rhabdomyosarcoma (RMS).

OUTLINE: Archived serum samples are analyzed for miR-206 expression.

PROJECTED ACCRUAL: A total of 15 samples from patients with alveolar rhabdomyosarcoma (RMS), 15 from patients with embryonal RMS, and 10 from patients without RMS will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Serum specimens of rhabdomyosarcoma (RMS), embryonal RMS, and non-RMS available from the Soft Tissue Sarcoma committee of Children's Oncology Group

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rhabdomyosarcoma (RMS), embryonal RMS, and non-RMS.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serum miR-206 as a biomarker for RMS

CONTACTS AND LOCATIONS:
Overall Officials: Hajime Hosoi, MD, Principal Investigator — Kyoto Prefectural University of Medicine